CLINICAL TRIAL: NCT00591747
Title: Strength Training for Older Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1836; 050106
Record Dates: First submitted 2007-12-31; First posted 2008-01-11 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Breast Neoplasm; Osteoporosis, Postmenopausal
Keywords: randomized clinical trial; elderly; cancer survivor; bone health; body composition; signs and symptoms
MeSH Terms: conditions — Breast Neoplasms; Osteoporosis, Postmenopausal; Signs and Symptoms | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Progressive resistance training program 3 times a week for 12 months
  Interventions: Behavioral: Resistance Exercise
- 2 (Active Comparator): Flexibility training 3 times a week for 12 months
  Interventions: Behavioral: Flexibility Training

INTERVENTIONS:
Behavioral: Resistance Exercise — 60 minute sessions 3 times a week of moderate-vigorous lower and upper body free-weight strength training plus impact training (jumps). Two of the three sessions are conducted in a supervised setting at a university fitness facility and the third session is a modified version of the exercise program performed at home. Participants are in the exercise program for 12 months
  Arms: 1
Behavioral: Flexibility Training — 60 minute session 3 times a week focusing on whole body flexibility (stretching) and relaxation (progressive neuromuscular relaxation, focused breathing) exercises. Exercises are selected to be non-weight bearing and require minimal muscle strength in order to provide a contrast to the intervention arm. Two sessions are conducted in a supervised setting at a university fitness center and the third is a home-based version of the program performed at home.
  Arms: 2

SUMMARY:
Women aged 50 and older are disproportionately affected by breast cancer, not only in terms of new diagnoses, but also in terms of survivorship. Approximately 85% of women who receive a first diagnosis of breast cancer are aged 50 and over, thus older women constitute the largest group of breast cancer survivors. Yet, few studies have focused on evaluating whether physical activity and exercise interventions affect long-term symptoms, physical fitness and function, and body composition of older breast cancer survivors. Due to the combined effects of breast cancer, related treatments and aging it is likely that exercise is even more beneficial for older breast cancer survivors than for younger survivors. Along with the cancer-related symptom of fatigue common to cancer survivors, older survivors face age-related declines in bone and muscle mass, muscle strength, bone health and physical function (gait and balance) that are likely exacerbated by reduced physical activity in survivorship and side effects of adjuvant cancer treatment. All women, regardless of age, are at risk for breast cancer recurrence. Recent epidemiologic evidence suggests a link between exercise and reduced risk of cancer recurrence in breast cancer survivors. Strength training is specifically suited to reverse or slow age-related declines in bone, muscle, strength and function and has shown promise to reduce cancer-related fatigue. However, no controlled trials of strength training in older breast cancer survivors have been conducted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with early stage breast cancer at age of 50 or older
* Completed adjuvant therapy, radiation +/- chemotherapy but selective estrogen receptor modulators (SERMS), (aromatase inhibitors (AIs) ok) at least 1 year prior to enrollment

Exclusion Criteria:

* Cognitive difficulties that preclude answering the survey questions, participating in performance testing or giving informed consent
* Diagnosed osteoporosis
* Current regular participation in planned impact activities or resistance training (more than 2 times a week for 30 minutes at a time)
* Medication that contraindicates participation in moderate intensity strength training or previous use of medications known to affect bone metabolism
* Movement or neurologic disorder, not including chemo-induced peripheral neuropathy

Ages: 50 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2005-11; Primary Completion 2009-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Physical functioning (muscle strength, gait and balance), self-report physical and mental health, and fatigue | 12 months

SECONDARY OUTCOMES:
Body composition (fat mass, muscle mass) and bone mineral density of the lumbar spine and proximal femur | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kerri M Winters, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU School of Nursing, Portland, Oregon, United States

REFERENCES:
- [Result] Winters-Stone KM, Dobek J, Nail L, Bennett JA, Leo MC, Naik A, Schwartz A. Strength training stops bone loss and builds muscle in postmenopausal breast cancer survivors: a randomized, controlled trial. Breast Cancer Res Treat. 2011 Jun;127(2):447-56. doi: 10.1007/s10549-011-1444-z. Epub 2011 Mar 19. PMID 21424279
- [Result] Winters-Stone KM, Dobek J, Bennett JA, Nail LM, Leo MC, Schwartz A. The effect of resistance training on muscle strength and physical function in older, postmenopausal breast cancer survivors: a randomized controlled trial. J Cancer Surviv. 2012 Jun;6(2):189-99. doi: 10.1007/s11764-011-0210-x. Epub 2011 Dec 23. PMID 22193780
- [Result] Dobek J, Winters-Stone KM, Bennett JA, Nail L. Musculoskeletal changes after 1 year of exercise in older breast cancer survivors. J Cancer Surviv. 2014 Jun;8(2):304-11. doi: 10.1007/s11764-013-0313-7. Epub 2013 Dec 7. PMID 24317968
- [Result] Winters-Stone KM, Leo MC, Schwartz A. Exercise effects on hip bone mineral density in older, post-menopausal breast cancer survivors are age dependent. Arch Osteoporos. 2012;7(1-2):301-6. doi: 10.1007/s11657-012-0071-6. Epub 2012 Mar 20. PMID 23225299
- [Derived] Ernst M, Wagner C, Oeser A, Messer S, Wender A, Cryns N, Brockelmann PJ, Holtkamp U, Baumann FT, Wiskemann J, Monsef I, Scherer RW, Mishra SI, Skoetz N. Resistance training for fatigue in people with cancer. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD015518. doi: 10.1002/14651858.CD015518. PMID 39606939
- [Derived] Winters-Stone KM, Wood LJ, Stoyles S, Dieckmann NF. The Effects of Resistance Exercise on Biomarkers of Breast Cancer Prognosis: A Pooled Analysis of Three Randomized Trials. Cancer Epidemiol Biomarkers Prev. 2018 Feb;27(2):146-153. doi: 10.1158/1055-9965.EPI-17-0766. Epub 2017 Nov 15. PMID 29141853